CLINICAL TRIAL: NCT00866424
Title: A Prospective Study on Efficacy of Hyperbaric Oxygenation Treatment for Patients With Trigeminal Neuralgia: a Randomized, Double-Blind, Mock Hyperbaric Chamber -Controlled, Parallel-Group Trial
Brief Title: Clinical Trial of Hyperbaric Oxygen Treatment in Trigeminal Neuralgia Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Lize Xiong/A Prospective Study on Efficacy of Hyperbaric Oxygenation Treatment for Patients with Trigeminal Neuralgia: a Randomized, Double-blind, Mock hyperbaric Chamber -Controlled, Parallel-Group Trial, Fourth Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20080327-1
Record Dates: First submitted 2009-01-14; First posted 2009-03-20 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-01

CONDITIONS: Trigeminal Neuralgia; Pain
Keywords: trigeminal neuralgia; pain; HBO; VAS; MGPQ
MeSH Terms: conditions — Trigeminal Neuralgia; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A,2, II (Experimental)
  Interventions: Procedure: Hyperbaric oxygen, Mock hyperbaric chamber

INTERVENTIONS:
Procedure: Hyperbaric oxygen, Mock hyperbaric chamber — Hyperbaric oxygen treatment for 10 days in treatment groups and mock hyperbaric chamber treatment for 10 days in control groups.
  Hyperbaric oxygen treatment: While in the hyperbaric chamber the subjects breathe 100% oxygen saturation with mask at 2.0bars.
  Mock hyperbaric chamber treatment: The subjects breathe air freely in the imitation environment chamber at 1.0bars.
  Other Names: the delivery of oxygen in a pressurised chamber

SUMMARY:
The purpose of this study is to determine whether the hyperbaric oxygen treatment reduces pain and improve the life quality in trigeminal neuralgia patients.

DETAILED DESCRIPTION:
Trigeminal neuralgia(TN) is a recurrent severe shooting neuropathic pain. Treatment of this pain continues to be a challenge in clinical pain management. Hyperbaric oxygen (HBO) has been used of neuropathic diseases, which can improve blood partial pressure of oxygen, reduce edema, relieve neural oppression and attenuate inflammatory response. The hypothesis of this protocol is that hyperbaric oxygen treatment could relieve neuropathic pain and improve the quality of life in TN patients. Visual analogue scale (VAS) and the mcgill pain questionnaire (MGPQ) will be assessed before the initiation of the study, after hyperbaric oxygen (HBO) treatment and at monthly intervals for the subsequent 3 months. Titration of dosage and pain frequency will be recorded throughout the study. Clinical global impression (CGI) by the individual patient will be evaluated at monthly intervals after HBO treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70
2. Primary TN patient (MRI examination support diagnosis)
3. Suffering from this pain for at least 3 months
4. VAS﹥40mm
5. Patient can assess pain intensity correctly

Exclusion Criteria:

1. Undergone surgery for TN(including nerve injections) within the last year
2. Oral medicine change within the last week
3. With other diseases of nervous system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-01 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
visual analogue scales (VAS), the mcgill pain questionnaire (MGPQ). | after HBO treatment

SECONDARY OUTCOMES:
visual analogue scales (VAS), the mcgill pain questionnaire (MGPQ),pain frequency, titration of dosage, clinical global impression (CGI) | at monthly intervals for the subsequent 6 after hyperbaric oxygen (HBO) treatment

CONTACTS AND LOCATIONS:
Overall Officials: Li ze Xiong, MD, Study Chair — Xijing Hospital, Fourth Military, Medical Univercity
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China